CLINICAL TRIAL: NCT01950533
Title: The Utility of Food-Specific IgE Measured With the IMMULITE 2000 Assay to Predict Symptomatic Food Allergy
Acronym: IMMULITE 2000
Status: Completed | Type: Observational
Sponsor: National Jewish Health (Other)
Responsible Party: Sponsor
Other Study IDs: IMMULITE 2000; Siemens (Other: Siemens)
Record Dates: First submitted 2013-09-23; First posted 2013-09-25 (Estimated); Last update posted 2020-10-19 (Actual); Status verified 2020-10

CONDITIONS: Peanut Allergy; Milk Allergy; Egg Allergy
Keywords: Peanut allergy; Milk allergy; Egg allergy; Pediatric; Adult; Food allergy
MeSH Terms: conditions — Peanut Hypersensitivity; Milk Hypersensitivity; Egg Hypersensitivity; Food Hypersensitivity

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (3):
- Peanut allergic: Subjects allergic to peanuts by oral food challenge
  Interventions: Procedure: Oral food challenge
- Milk allergic: Subjects allergic to milk by oral food challenge
  Interventions: Procedure: Oral food challenge
- Egg allergic: Subjects allergic to egg by oral food challenge
  Interventions: Procedure: Oral food challenge

INTERVENTIONS:
Procedure: Oral food challenge — Confirmation of allergy to egg, milk and/or peanut through an oral food challenge or documentation of a positive oral food challenge.

SUMMARY:
Food allergy is on the rise within the pediatric population. Having food allergy can cause medical, nutritional and psychological issues in those who suffer with it. Although making the appropriate diagnosis of food allergy is very important, properly diagnosing food allergy has been a challenge. Skin prick testing and food-specific IgE testing of the blood can give positive results that are false. Currently, Oral Food Challenges are the best way to diagnose a food allergy. Unfortunately, Oral Food Challenges are time consuming and may not be readily available to suspected food allergy sufferers. This study is designed to examine the effectiveness of an allergy-detecting blood test called IMMULITE 2000 manufactured by the study sponsor, Siemens.

ELIGIBILITY:
Inclusion Criteria:

* Age 3 to 21 years of either sex and any race
* Physician-diagnosed food allergy or convincing clinical history of food allergy to milk, egg, and/or peanut AND a Skin prick test positive to milk, egg, and/or peanut (diameter of wheal > 3 mm or greater than negative control) orOR a detectable serum food-specific IgE level (ImmunoCAP and/or IMMULITE > 0.35 kUA/L) to milk, egg, and/or peanut
* If no history of clinical reactivity to milk, egg, or peanut, then a positive skin prick test to milk, egg, and/or peanut (diameter of wheal > 3 mm or greater than negative control) OR a detectable serum food-specific IgE level within the previous 4 months to milk, egg, and/or peanut
* Written informed consent from parent/guardian and assent (when age appropriate).
* Willingness to submit specimen for laboratory serum IgE testing

Exclusion Criteria:

* Inability to discontinue antihistamines for skin prick testing and OFCs
* Current allergy to placebo ingredient (oat flour) OR reaction to any dose of placebo at the qualifying OFC
* FEV1 value <80% predicted OR any clinical features of moderate or severe persistent asthma, as defined by the 2007 NHLBI guidelines table for classifying asthma baseline severity (Step 3 or above), at the time of entry into the study
* Use of , and >high medium daily doses of inhaled corticosteroids, as defined by the 2007 NHLBI guidelines inhaled corticosteroid dosing table (500500 μg/day fluticasone or equivalents for an adult) or a long acting beta-agonist (LABA) to control asthma.
* Asthma requiring either:

> 1 hospitalization in the past year for asthma or > 1 ER visit in the past 6 months for asthma

* History of intubation due to allergies or asthma
* Use of steroid medications (IV, IM or oral) for asthma in the following manners:

  * history of daily oral steroid dosing for >1 month during the past year or
  * burst or steroid course/burst in the past 3 months or
  * >2 burst oral steroid courses/bursts in the past year
* History of intubation due to allergies or asthma
* Life-threatening allergic reaction (e.gi.e., respiratory compromise, hypoxia, hypotension, use of epinephrine) to study food(s) (e.g., milk, egg, and/or peanut) within last 1 year
* Diagnosis of active eosinophilic gastrointestinal disease in the past year
* Severe or poorly controlled atopic dermatitis, as assessed by a three-item severity (TIS) score of 6 or greater (see Appendix I)
* Use of omalizumab or other non-traditional forms of allergen immunotherapy (e.g., oral or sublingual), immunomodulatory therapy (not including corticosteroids), or biologic therapy within the past year
* Uncontrolled hypertension
* Any use of β-blockers (oral), angiotensin-converting enzyme (ACE) inhibitors, angiotensin-receptor blockers (ARB) or calcium channel blockers
* Other significant medical conditions (e.g., liver, gastrointestinal, kidney, cardiovascular, pulmonary disease, or blood disorders), which, in the opinion of the Investigator, make the subject unsuitable for induction of food reactions
* Pregnancy

Ages: 3 Years to 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Study population will be primarily obtained from the pediatric clinic at National Jewish Health from those suspected of egg, milk and/or peanut food allergy.
Sampling Method: Non-Probability Sample
Enrollment: 102 (Actual)
Dates: Start 2013-09 (Actual); Primary Completion 2017-03-29 (Actual); Study Completion 2017-03-29 (Actual)

PRIMARY OUTCOMES:
Relationship between food specific IgEs | approximately 2 weeks
  To determine the relationship between food-specific IgE to whole proteins of milk, egg, and peanut using the IMMULITE 2000 assay and OFC outcomes.

SECONDARY OUTCOMES:
Logisitic regression analyses on data | approximately 2 weeks
  To compare the results of logistic regression analyses using the IMMULITE 2000 assay and food challenge outcome data to data obtained in parallel using the ImmunoCAP assay for food-specific IgE antibodies.

CONTACTS AND LOCATIONS:
Overall Officials: Erwin Gelfand, MD, Principal Investigator — National Jewish Health
Locations (1):
- National Jewish Health, Denver, Colorado, United States